CLINICAL TRIAL: NCT00734617
Title: Concurrent Nicotine Patch / Denicotinized Cigarette Therapy for Smoking Cessation II
Acronym: CON NIC II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00001223
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Results first posted 2011-03-01 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2011-02

CONDITIONS: Cigarette Smoking
Keywords: Cigarette; Nicotine
MeSH Terms: conditions — Cigarette Smoking | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Less Dependent Smokers (Experimental)
  Interventions: Drug: Nicotine Patch
- More Dependent Smokers (Experimental)
  Interventions: Drug: Nicotine Patch

INTERVENTIONS:
Drug: Nicotine Patch — Groups 1 & 3 1-21mg Nicotine patch and 1-placebo for 2 wks pre quit day and 4 wks post quit day
  Groups 2 & 4 2-21mg Nicotine Patches for 2 wks pre quit day and 4 wks post quit day

SUMMARY:
The main goals of the study are to assess benefits of higher doses of the nicotine patch prior to smoking cessation for high- and low-dependent smokers, and to investigate the potential relationship between genetic factors and smoking cessation success. There will be a two-week double-blind pre-cessation exposure to nicotine patch treatment in a sample of 240 high-dependent & 240 low-dependent smokers; half of each group will wear two 21mg nicotine patches (42mg) daily, and half will wear one 21mg nicotine patch and one comparable placebo patch daily, resulting in the following four conditions (120 subjects each) during the 2-week pre-quit period: 1) Less Dependent/21mg nic., 2) Less Dependent/42mg nic., 3) More Dependent/21mg nic., and 4) More Dependent/42mg nic. After the quit date, subjects will continue with the same nicotine dosage for the 1st 4 weeks; after that the treatment will no longer be double-blind as only nicotine patches will be used: all subjects will wear one 21-mg patch daily for 2 weeks, one 14-mg patch daily for the following 2 weeks, and one 7-mg patch for the remaining 2 weeks. The four treatment groups will be distributed over 4 sites: Durham, Raleigh, Charlotte, and Winston-Salem. After the screening visit, subjects will have 7 lab visits: at 2 weeks, 1 week, and 1 day prior to the quit-smoking date, and at 1 week, 3 weeks, 6 weeks and 10 weeks after the quit-smoking date.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18-65 years old, have smoked an average of at least 10 cigarettes per day for three cumulative or continuous years of a brand that delivers (by Federal Trade Commission rated yields) at least 0.5 mg nicotine, have an expired air carbon monoxide reading of at least 10 ppm, and express a desire to quit smoking. Additionally, subjects must express a willingness to switch to denicotinized cigarettes. A more dependent smoker is defined as someone with an FTND score of seven or greater. A less dependent smoker is defined as someone with an FTND score of less than seven.

Exclusion Criteria:

* For those with a known history of hypertension, systolic >140 mm Hg, diastolic >100 mm Hg); hypotension (systolic <90 mm Hg, diastolic <60 mm Hg) Participants with hypertension or hypotension may, however, be allowed to participate in the study if the study physician or P.A. determines that the condition is stable, controlled by medication, and in no way jeopardizes the individual's safety. Subjects with no previous diagnosis of hypertension may have a screening blood pressure up to 160/100. Potential subjects who report coronary heart disease; heart attack; cardiac rhythm disorder (irregular heart rhythm); chest pains (unless history, exam, and EKG clearly indicate a non-cardiac source); cardiac (heart) disorder (including but not limited to valvular heart disease, heart murmur, heart failure); history of skin allergy; active skin condition (psoriasis) within the last five years; skin disorder except minor skin conditions (including but not limited to facial acne, minor localized infections, and superficial minor wounds.); liver or kidney disorder (except kidney stones, gallstones); gastrointestinal problems or disease other than gastroesophageal reflux or heartburn; ulcers; lung disorder (including but not limited to COPD, emphysema, and asthma); brain abnormality (including but not limited to, stroke, brain tumor, seizure disorder); history of fainting; problems giving blood samples; difficulty passing urine; diabetes treated with insulin, non-insulin treated diabetes (unless glucose is less than 180mg/dcl and HbA1c is less than 7%); current cancer or treatment for cancer in the past 6 months(except basal or squamous cell skin cancer); other major medical condition; current psychiatric disease (with the exception of depression, anxiety disorders, OCD and ADHD) will be excluded from the study. Potential subjects who do not have a self reported diagnosis of the above listed conditions may be excluded if the study physician or P.A. determines that the history, physical findings, EKG, or laboratory studies reveal information that may jeopardize the subject's safe study participation.

Potential subjects who have abused alcohol or drugs, or have used within the last 30 days experimental (investigational) drugs, psychiatric medications (including antidepressants, anti-psychotics) or any other medications that are known to affect smoking cessation (e.g. clonidine) will be excluded. Potential subjects who have used smokeless tobacco (chewing tobacco, snuff), cigars, pipes, nicotine replacement therapy, or other smoking cessation treatment within the last 2 weeks will be excluded. Pregnant or nursing mothers will be excluded.

Use of non-opiate medications for pain or sleep will be allowed. For medical conditions that do not appear above, the study physician will be consulted and if the medical condition does not jeopardize safe study participation, then the subject may be enrolled.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 479 (Actual)
Dates: Start 2007-08; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jed E Rose, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Uhl GR, Drgon T, Johnson C, Ramoni MF, Behm FM, Rose JE. Genome-wide association for smoking cessation success in a trial of precessation nicotine replacement. Mol Med. 2010 Nov-Dec;16(11-12):513-26. doi: 10.2119/molmed.2010.00052. Epub 2010 Aug 24. PMID 20811658
- [Derived] Rose JE, Behm FM, Drgon T, Johnson C, Uhl GR. Personalized smoking cessation: interactions between nicotine dose, dependence and quit-success genotype score. Mol Med. 2010 Jul-Aug;16(7-8):247-53. doi: 10.2119/molmed.2009.00159. Epub 2010 Mar 17. PMID 20379614

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment start date: 8/20/2007 Recruitment end date: 3/19/2008 Recruitment locations: Duke Center for Nicotine & Smoking Cessation Research offices located in Charlotte, Durham, Raleigh and Winston-Salem NC.
Pre-assignment Details: Participants were excluded for the following reasons:
  DID NOT MEET INCLUSION CRITERIA: 78 MET EXCLUSION CRITERIA: 74 UNABLE TO MEET STUDY REQUIREMENTS: 9 REFUSED TO PARTICIPATE: 18 LOST TO CONTACT (PRIOR TO V1): 30 LAB RESULTS: 64 MD/PA REFUSAL: 179 30 DAYS PAST PHYSICAL SCREENING: 1
Period: Overall Study
Arm/Group | Less Dependent | More Dependent
Started | 249 | 230
Completed | 142 | 128
Not Completed | 107 | 102
Not completed — Adverse Event | 4 | 7
Not completed — Withdrawal by Subject | 103 | 95

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Less Dependent | More Dependent | Total
Number analyzed (Participants) | 249 | 230 | 479
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 249 | 230 | 479
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (11.4) | 44.34 (10.92) | 43.53 (11.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 136 | 272
  Male | 113 | 94 | 207
Region of Enrollment [Number; unit: participants]
  United States | 249 | 230 | 479

OUTCOME MEASURES:

1. Primary Outcome: Continuous Abstinence From Smoking at Ten Weeks Post-quit
Description: Continuous abstinence from the target quit date through the end of treatment (10 weeks) was assessed based on self reports of continuous abstinence (i.e., no lapses) that were confirmed by end-expired CO levels ≤ 10 ppm.
Time Frame: May 2009
Measure: Number; unit: participants
Arm/Group | Less Dependent | More Dependent
Number analyzed (Participants) | 249 | 230
participants
  21mg Nicotine Patch | 31 | 21
  42mg Nicotine Patch | 17 | 26

ADVERSE EVENTS:
Arm/Group | Less Dependent | More Dependent
Serious Adverse Events (participants affected / at risk) | 0/249 | 0/230
Other Adverse Events (participants affected / at risk) | 0/249 | 0/230

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes